CLINICAL TRIAL: NCT02927197
Title: A Randomized, Controlled Study on the Effects of LearningRx Brain Training for Improving Cognitive Skills in Students Ages 8-14
Brief Title: LearningRx Brain Training for Children 8-14
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gibson Institute of Cognitive Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GICR-1005
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Learning Problems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LearningRx Cognitive Training (Experimental): The intervention is a 60-hour one-on-one cognitive training program
  Interventions: Behavioral: LearningRx cognitive training
- Waitlist Control (No Intervention): The treatment-as-usual control group will begin the intervention when the experimental arm has completed the intervention.

INTERVENTIONS:
Behavioral: LearningRx cognitive training — A clinician will deliver forty 90-minute cognitive training sessions over 12-14 weeks for a total of 60 training hours. There are 23 different categories of training procedures sequenced in intensity and difficulty for a total of more than 1000 training tasks.
  Other Names: ThinkRx
  Arms: LearningRx Cognitive Training

SUMMARY:
The purpose of this study is to examine changes in multiple cognitive skills after completing 60 hours of cognitive training with ThinkRx, a LearningRx program.

DETAILED DESCRIPTION:
In a two-phase randomized controlled study, investigators will examine the effects of a one-on-one cognitive training program on memory, visual and auditory processing, processing speed, reasoning, attention, and General Intellectual Ability (GIA) score for students ages 8-14. In Phase 1, participants will be randomly assigned to either an experimental group to complete 60 hours of one-on-one cognitive training or to a wait-list control group. In Phase 2, the wait-list control group will complete the intervention using an alternative delivery model: 50% clinician delivered and 50% digital delivery.

ELIGIBILITY:
Inclusion Criteria:

* Between 8-14 years of age, living in the greater Colorado Springs area, screening GIA score between 70 and 130

Exclusion Criteria:

* None

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Evidence of overall cognitive function improvement | within 14 days after completing the intervention
  Confirmed by pretest to post-test change on the Woodcock Johnson III - Tests of Cognitive Abilities (WJ III): General Intellectual Ability composite score

SECONDARY OUTCOMES:
Evidence of improvement in school performance | Within two years after completing the intervention
  Confirmed by improvement in school achievement tests and grade reports
Evidence of improvement in working memory | within 14 days after completing the intervention
  Confirmed by pretest to posttest change on the WJ III: Numbers Reversed test
Evidence of improvement in long-term memory | within 14 days after completing the intervention
  Confirmed by pretest to posttest change on the WJ III: Visual-Auditory Learning Delayed test
Evidence of improvement in fluid reasoning | within 14 days after completing the intervention
  Confirmed by pretest to posttest change on the WJ III: Concept Formation test
Evidence of improvement in processing speed | within 14 days after completing the intervention
  Confirmed by pretest to posttest change on the WJ III: Visual Matching test
Evidence of improvement in visual processing | within 14 days after completing the intervention
  Confirmed by pretest to posttest change on the WJ III: Spatial Relations test
Evidence of improvement in auditory processing | within 14 days after completing the intervention
  Confirmed by pretest to posttest change on the WJ III: Sound Blending test
Evidence of improvement in attention | within 14 days after completing the intervention
  Confirmed by pretest to posttest change on the National Institutes of Health (NIH) Cognition Toolbox attention test

CONTACTS AND LOCATIONS:
Overall Officials: Dick M Carpenter, PhD, Principal Investigator — University of Colorado, Colorado Springs
Locations (1):
- Gibson Institute of Cognitive Research, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Harvard Dataverse

REFERENCES:
- [Result] Carpenter DM, Ledbetter C, Moore AL. LearningRx Cognitive Training Effects in Children Ages 8-14: A Randomized Controlled Trial. Appl Cogn Psychol. 2016 Sep-Oct;30(5):815-826. doi: 10.1002/acp.3257. Epub 2016 Aug 2. PMID 27867257